CLINICAL TRIAL: NCT07400887
Title: Onderzoek Naar de Kennis Over en Houding Ten Opzichte Van Non-binaire Personen in Vlaanderen (Deel 1, Kwantitatief)
Brief Title: Knowledge About and Attitudes Towards Non-binary Persons in Flanders (Part 1: Quantitative Study)
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: IPSOS (Industry)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0115
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non-binary
Keywords: Online survey; Attitudes; Non-binary; Knowledge
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flemish participants: 1000 Flemish adult participants, randomly selected from Ipsos panel. No intervention.
- Dutch participants: 1000 Dutch adult participants, randomly selected from Ipsos panel. No intervention.

SUMMARY:
The goal of this observational study is to investigate the knowledge about and attitudes towards non-binary individuals in Flemish adults. The main questions it aims to answer are:

To which degree does the Flemish population have knowledge about non-binary persons? What are the attitudes of the Flemish population towards non-binary persons? What factors influence the attitudes towards non-binary persons? Furthermore, the aim is to create a survey to measure knowledge about and attitudes towards non-binary persons.

Participants will complete an online survey.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Living in Flanders or the Netherlands
* enrolled in Ipsos ISO-certified panel

Exclusion Criteria:

* 17 or <17 years old
* not living in Flanders or the Netherlands
* not enrolled in Ipsos ISO-certified panel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ipsos ISO-certified panel
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Attitudes towards non-binary persons | At the time of enrollment
  An online survey of 16 questions to measure attitudes was developed based on existing literature. A scale of 15 questions was then developed to make follow-up measurements possible.

SECONDARY OUTCOMES:
Knowledge about non-binarity | At the time of enrollment
  The online survey included questions asking about respondents' familiarity with the term "non-binary" and with non-binary persons, and about their definition of the concept

CONTACTS AND LOCATIONS:
Overall Officials: Joz Motmans, Principal Investigator — University Hospital, Ghent
Locations (1):
- Universitair Ziekenhuis Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.uzgent.be/nl/patient/zoek-een-arts-of-dienst/centrum-voor-seksuologie-en-gender/genderzorg/projecten-en-onderzoeken-centrum-voor-seksuologie-en-gender